CLINICAL TRIAL: NCT06790953
Title: Clinical Efficacy of Novel Biogenically Fabricated Titania Nanoparticles Enriched Mouth Wash in Treating the Tooth Dentine Hypersensitivity: a Randamized Clinical Trial
Brief Title: Efficacy of Novel Titania Nanoparticles Enriched Mouth Wash in Treating Dentine Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Afsheen Mansoor, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOD/ERB/2024/36-200
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Dentine Hypersensitivity
Keywords: Bacillus coagulans; Biogenic; Dentin Hypersensitivity; Nanoparticles; Titanium oxide (TiO2 Nps)
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: In this study, participants will be allocated in two groups by Consecutive random sampling technique
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This is a triple-blinded study in which the participant, care provider and outcome assessor will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-A: Conventional Mouth wash . (Experimental): Group A will receive conventional mouthwash for treatment of dentin hypersensitivity
  Interventions: Procedure: Group- A Conventional Sensed Mouth Wash
- Group-B: Novel Titania nanoparticles Mouth wash (Experimental): Group B will receive novel Titania nano particles reinforced mouthwash for treatment of dentin hypersensitivity
  Interventions: Procedure: Group-B Novel Titania nanoparticles enriched Mouth Wash

INTERVENTIONS:
Procedure: Group- A Conventional Sensed Mouth Wash — In Group- A Conventional Sensed Mouth Wash will be used for treatment of Dentin hypersensitivity.
  Visual Analogue scoring system will be used to calculate the dentin hypersensitivity.
  Arms: Group-A: Conventional Mouth wash .
Procedure: Group-B Novel Titania nanoparticles enriched Mouth Wash — In Group-B Novel Titania nanoparticles enriched Mouth wash will be used to treat the Dentin hypersensitivity.
  Visual Analogue scoring system will be used to calculate the dentin hypersensitivity.
  Arms: Group-B: Novel Titania nanoparticles Mouth wash

SUMMARY:
Randomized Clinical trial to compare the reduction in dentin hypersensitivity after incorporating biogenically fabricated titania nanoparticles enriched Mouth Wash and Conventional Mouth Wash.Participants ranging between 20-50 years were allocated in two groups. Group A will use Conventional Mouth Wash without Nanoparticles. Group B will use titania nanoparticles enriched Mouth Wash. Both will use them for three months and then their VAS scoring will be checked.

DETAILED DESCRIPTION:
In this study Novel biogenically fabricated titania nanoparticle reinforced Mouth Wash will be evaluated for dentine sensitivity . Participants following Inclusion criteria will be allocated in this study by Consecutive random sampling technique. Participants will be divided into two groups i.e Group-A and Group-B with dentin sensitivity of 30-80. Group A will be given Conventional Mouth Wash for three months and Group-B will be given titania nanoparticles enriched Mouth Wash for three months for the sensitivity. Sensitivity will be assessed using Visual analog scale (VAS) mean score after 1 month and then three months.

ELIGIBILITY:
Inclusion Criteria:

* Participants ranging between 20-50 years, good general health but developed dentine sensitivity associated with tooth surface wear and loss during the past 6 months.
* There was no history of allergy.
* Participants did not use any mouth wash , dentifrice or medication in the last 3 months.
* The involved teeth were viable, non-shaky, devoid of any decay, cracks and fillings.
* There was an essential positive response to the provoking Air stimuli.
* These teeth should display the visible signs of tooth loss and wear such as : attrition, abrasion, erosion and abfraction.

Exclusion Criteria:

* Participants that might have developed allergy or used medications during the last 2 weeks or more.
* The teeth having cracks, decay and fillings were also excluded. Patients who have undergone any periodontal surgery or gross periodontal issues.
* Participants who used any desensitisizing toothpastes/mouthwashes and tooth bleaching agents within 2 months of the trial were also excluded positively.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Post mouth wash utilization Dentine Hypersensitivity | 3 months
  Evaluation of dentine hypersensitivity with Conventional Mouth Wash without titania nanoparticles and Novel Nps Mouth Wash with titania nanoparticles on human tooth dentin. Visual analog scale with scoring from 0 to 100 where Score 100 means worst outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Afsheen Mansoor, PhD, Principal Investigator — School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad.
Locations (1):
- School of Dentistry, Pakistan Institute of Medical Sciences, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboelenein AZ, Riad MI, Haridy MF. Effect of a Self-Etch Adhesive Containing Nanobioglass on Postoperative Sensitivity of Posterior Composite Restorations - A Randomized Trial. Open Access Maced J Med Sci. 2019 Jul 25;7(14):2313-2320. doi: 10.3889/oamjms.2019.585. eCollection 2019 Jul 30. PMID 31592280